CLINICAL TRIAL: NCT05008289
Title: Effects of Magnetic Stimulation of the Dorsal Spinal Cord on Gait in Patients With Parkinson´s Disease and Deep Brain Stimulation
Acronym: TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16233819800000068
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; magnetic transcutaneous stimulation; spinal cord stimulation; gait in parkinson disease; deep brain stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACTIVE (Active Comparator): Magnetic transcutaneous spinal cord stimulation
  Interventions: Device: Magnetic transcutaneous spinal cord stimulation; Device: Transcutaneous electrical nerve stimulation
- PLACEBO (Sham Comparator)
  Interventions: Device: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: Magnetic transcutaneous spinal cord stimulation — In the active group, non-invasive spinal cord stimulation will be applied by placing a circular magnetic coil (Magventure®️ MagPro®️ R20) on the skin, in the upper thoracic region (thoracic level T2-T3). The intensity of stimulation will represent 100% of the motor threshold, which is determined by abdominal muscle contractions, found from single pulses, gradually applied every 10 seconds until the onset of contractions. The intermittent theta burst stimulation protocol will consist of 20 stimulation trains, with an interval of 8 seconds between trains, each train will have 20 bursts, and each burst will have 3 pulses at 50 Hertz repeated at 5 Hertz. In total 1200 pulses will be applied for 3 minutes and 58 seconds.
  Other Names: TMS
  Arms: ACTIVE
Device: Transcutaneous electrical nerve stimulation — To create a sensation of muscle contraction and impression of active stimulation, both the placebo and active groups will be subjected to the sensory effect of transcutaneous electrical neurostimulation (TENS). The surface electrodes of TENS (model Neurodyn®️, Ibramed®️) will be placed in parallel at the height of the thoracic level T2-T3, with the following parameters: 80Hertz, 150ms, approximately at 60 miliampère.
  In the placebo group, a coil will be allocated in the thoracic region T2-T3, however this coil will not be connected to the stimulation device, and another active coil will be positioned about 15cm behind, away from its field of view, to provide the idea from the sound stimulus that it is being stimulated.
  Other Names: TENS

SUMMARY:
Gait disorders are symptoms that significantly compromise the quality of life and functionality of patients with Parkinson's disease (PD). When they are not responsive to drug dopaminergic therapy and deep brain stimulation (DBS), the management of these symptoms is a challenge in clinical practice. Although deep brain stimulation is useful in the motor symptoms of Parkinson's disease, gait symptoms remains a challenge in patients undergoing this therapy. This is because, in addition to adjustments in the DBS programming not adding evident benefit in some patients with gait disorders, motor symptoms tend to progress over the years. In this context, spinal cord invasive electrical stimulation was proposed as a potential and effective therapy in a group of patients with PD who presented with gait impairment. More recently, the application of transcutaneous magnetic stimulation of the spinal cord has emerged as a possible therapeutic option, as it could stimulate neural elements in a non-invasive way. The general objective will be to study the effect of transcutaneous magnetic stimulation of the spinal cord on gait in PD patients with deep brain stimulation refractory to dopaminergic therapy. The method of the present study will be a randomized, double-blind, placebo-controlled, parallel, phase II clinical trial that will evaluate the efficacy of transcutaneous magnetic stimulation of the spinal cord in patients with PD and deep brain stimulation who present gait disorders refractory to dopaminergic therapy. The primary outcome will be the change in gait speed between pre-stimulation and post-stimulation conditions between the two groups (active and placebo) assessed using the Timed Up and Go Test (TUG). Secondary outcomes will be the effects of stimulation on other gait measures (speed, step length, stride length, cadence, step width, sway time, support time and the presence of blocks), other motor symptoms (Unified Parkinson's Disease Rating Scale), cognitive alterations, quality of life and side effects. Statistical analysis will be performed using ANOVA for repeated measures and 38 patients will be included. The expected results are supported by transcutaneous magnetic stimulation of the spinal cord, which may improve gait disorders in participants with PD and DBS.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (non-pregnant) aged between 21 and 80 years;
2. Presence of deep brain stimulation in the subthalamic nucleus or globus pallidus
3. Participants with idiopathic Parkinson's disease at Hoehn Yahr stages between 2 and 4 during off-medication, whose primary symptom includes altered gait and/or balance (score equal to or greater than 1 on sub-item 2.12 of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) ["gait and balance"]). Patients should present the above symptoms even though they are optimized from a drug point of view and with optimized programming. The criteria to be optimized will be defined by a neurologist specialized in movement disorders who will evaluate the case.
4. Able to give informed consent in accordance with institutional policies;
5. Able to meet all testing and follow-up requirements as defined by the study protocol

Exclusion Criteria:

1. Patients with unstabilized psychiatric comorbidities;
2. Impossibility to consent to their participation in the study;
3. Patients with uncontrolled infection or other uncontrolled pre-existing medical conditions (eg, decompensated diabetes, high blood pressure, symptomatic pneumo or heart disease);
4. Concurrent treatment with other experimental drugs;
5. Pregnant or breastfeeding women;
6. Patients who cannot walk, not even with unilateral aid of a walking aid device or another person, when they are without their medication for Parkinson's Disease (off-medication);
7. Presence of cardiac pacemaker.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go - Test 5 Meters (TUG-Test 5M) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation
  The primary outcome will be the change in gait speed between pre-stimulation and post-stimulation conditions between the two groups (active and placebo) assessed using the 5-meter total Timed Up and Go Test (TUG). Mixel model ANOVA, with TUG as the dependent variable, and time and group as independent variables - "group" would have two levels ("active" and "placebo"). Our alternative hypotesis is that "the time vs. group" interaction effect is significant. Then we should use post hoc statistical tests to explore our data further and to compare the effects of active versus placebo at different time levels.

SECONDARY OUTCOMES:
Freezing of gait score (FOG SCORE) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in FOG SCORE between pre-stimulation and post-stimulation conditions.Minimum value 0 and maximum value 36. Higher value is worse.
Percentage of freezing by video analysis of Timed Up and Go - Test | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in percentage between pre-stimulation and post-stimulation conditions
Unified Parkinson's Disease Rating Scale (MDS-UPDRS) - Part III | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in UPDRS PART III between pre-stimulation and post-stimulation conditions. Minimum value 0 and maximum value 132. Higher value is worse.
Timed Up and Go - Test 5 Meters (TUG-Test 5M) Dual Task | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in gait speed between pre-stimulation and post-stimulation conditions
Mini Balance Evaluation Systems Test (Mini-BESTest) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in balance between pre-stimulation and post-stimulation conditions. Minimum value 0 and maximum value 108. Higher value is better.
New Freezing of Gait Questionnaire (NFOG-Q) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, fourteen days after the stimulation, twenty-one days after the stimulation, twenty-eight, thirty-five and forty-two days after the stimulation.
  Change in NFOG-Q between pre-stimulation and post-stimulation conditions. Minimum 0 Maximum 28. Higher value is worse.
Subitems 2.12 and 2.13 of Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, fourteen days after the stimulation, twenty-one days after the stimulation, twenty-eight, thirty-five and forty-two days after the stimulation
  Change between pre-stimulation and post-stimulation conditions
Parkinson's Disease Questionnaire 39 (PDQ-39); | Baseline, seven days after the stimulation, twenty-eight days after stimulation.
  Change in PDQ-39 between pre-stimulation and post-stimulation conditions. Minimum value 0% and maximum value 100%. Higher value is worse.
Falls Efficacy Scale (FES-I) | Baseline, seven days after the stimulation, twenty-eight days after stimulation.
  Change in FES-I between pre-stimulation and post-stimulation conditions. Minimum value 16 and maximum value 64. Higher value is worse.
Activities-specific Balance Confidence (ABC) Scale | Baseline, seven days after the stimulation, twenty-eight days after stimulation.
  Change in ABC scale between pre-stimulation and post-stimulation conditions. Minimum value 0 and maximum value 100%. Higher value is better.
Visual analog scale (VAS) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in pain between pre-stimulation and post-stimulation conditions. Minimum value 0 and maximum value 10. Higher value is worse.
Patient Global Impression of Change (PGIC) | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, fourteen days after the stimulation, twenty-one days after the stimulation, twenty-eight, thirty-five and forty-two days after the stimulation
  Impression of change post-stimulation conditions
Frontal assessment battery (FAB); | Baseline, immediately after the fifth day of stimulation, seven days after the stimulation, twenty-eight days after stimulation.
  Change in executive function between pre-stimulation and post-stimulation conditions. Minimum value 0 and maximum value 18. Higher value is better.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil